CLINICAL TRIAL: NCT07163962
Title: Maternal, Milk and Baby Markers of Group B Vitamin Metabolism in (Very) Preterm Infants at the Time of Discharge Home
Brief Title: THE B-BABIES STUDY: An Observational Study of Group B Vitamins in Preterm Infants
Acronym: B-BABIES
Status: Not yet recruiting | Type: Observational
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: Quadram Institute Bioscience (Other)
Responsible Party: Sponsor
Other Study IDs: 2024GRANT058
Record Dates: First submitted 2025-06-11; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Vitamin B-12 Deficiency
Keywords: Preterm infant; vitamin B12; Folate; Folic acid; Vitamin deficiency; Micronutrition
MeSH Terms: conditions — Vitamin B 12 Deficiency; Premature Birth; Avitaminosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, stool, urine, milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infancy may be associated with a risk of micronutrient depletion due to the high demands of rapid growth. This is particularly true when preterm birth occurs, as the period before term exhibits the highest rate of bodily growth across the lifespan. Folate and vitamin B12 are essential in development, and preterm infants may be particularly susceptible to deficiencies. This is the result of a combination of low stores and high requirements for fast growth and rapid red blood cell production in the context of multifactorial anaemia of prematurity. Micronutrient supply, including vitamin B12 and folate, is delivered through nutritional support, in the shape of parenteral nutrition, fortification of human milk of use of artificial formula. Most of this supplementation will be interrupted by the time the infant is getting ready for discharge home. The investigators previously reported high levels of serum folate in preterm infants at the time of discharge home and in early infancy, but there are no contemporary studies investigating the vitamin B12/folate status in this population. The investigators aim to investigate the prevalence of vitamin B12 deficiency in preterm infants at the time of discharge home.

DETAILED DESCRIPTION:
This is an observational, cross-sectional study of infants born preterm (gestational age at birth <37 weeks) and their mothers. The investigators aim to estimate the prevalence of vitamin B12 deficiency (low vitamin B12, high homocysteine and high MMA) under current nutritional guidelines in preterm (born <37 weeks) babies at the time of discharge in preterm infants under current nutritional guidelines.

The investigators will also study whether the risk of deficiency is different in those on an exclusive breast milk diet or in specific gestational age groups (late -34-36 weeks-, moderate -32-33 weeks-, very -28-32 weeks- and extremely -<28 weeks - preterm infants). Folate status will also be analysed. Exploratory outcomes include correlations between calculated intakes and vitamin levels, blood concentrations of other vitamins and cofactors in the same metabolic pathways, content of B vitamins in preterm maternal milk and performance of potential urinary markers of vitamin B12 deficiency in preterm infants.

The trial will take place in a single tertiary-level Neonatal Intensive Care Unit (NICU) and participant families will be recruited while their infant is an inpatient. The project has received Ethical Approval and Informed Consent for mother and baby/ies will be sought before participation.

This trial focuses on the population of preterm-born (<37 weeks of gestation) infants admitted to the Neonatal Unit.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth <37 weeks.
* Admission to one of the participating units.
* Full enteral milk feeds established by suck/nasogastric tube

Exclusion Criteria:

* Known or suspected chromosomal, genetic or metabolic abnormalities.
* Major congenital malformations
* Any intercurrent condition that precludes implementation of standard feeding protocols and requires specialized formulas or changes in standard vitamin supplementation.
* Any intercurrent condition that will interfere with the interpretation of results (renal impairment and hypothyroidism can lead to elevated tHcy and MMA, for example).

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants (born <37 weeks of gestation)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of biochemical vitamin B12 deficiency | between 34 and 44 weeks postmenstrual age, at the time of hospital discharge
  : Percentage of preterm infants with:
  * plasma cobalamin < 148 pmol/L.
  * MMA concentrations >0.26 µmol/L.
  * cB12 < -0.5.

SECONDARY OUTCOMES:
Prevalence of biochemical vitamin B12 deficiency in each gestational age group: late (34-36 weeks at birth), moderate (32-33 weeks at birth), very (28-32 weeks at birth) and extremely (<28 weeks at birth) preterm infants at the time of hospital discharge | between 34 and 44 weeks postmenstrual age, at the time of hospital discharge
  * Prevalence of folate deficiency (folate <10 nmol/L)/ elevated serum folate concentrations (>45.3 nmol/L) in preterm infants pre-discharge.
  * Quantification of UnMetabolized Folic Acid (UMFA) levels pre-discharge in preterm infants who receive any form of extra folic acid supplementation.

OTHER OUTCOMES:
To explore levels of other metabolites related to B12/folate pathways in preterm infants (including vitamin B6 and copper/zinc). | between 34 and 44 weeks postmenstrual age, at the time of hospital discharge
  Blood concentrations of vitamins B1, B2 and B6 (assessed by plasma levels of thiamine pyrophosphate, flavin adenine dinucleotide and pyridoxal 5'-phosphate, respectively).
Explore levels of B vitamins in human milk of mothers delivering prematurely | between 34 and 44 weeks postmenstrual age, at the time of hospital discharge
  Measurement of B1, B2, B6, folate and B12 in milk of mothers delivering prematurely. Correlations between concentration in breast milk and calculated total vitamin intake and infant blood levels will be also explored.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Isabel Iglesias-Platas, Principal Investigator — Norfolk and Norwich University Hospitals NHS Foundation Trust
Locations (1):
- Norfolk and Norwich University Hospital NHS Foundation Trust, Norwich, United Kingdom